CLINICAL TRIAL: NCT00748579
Title: A Phase II Open-Label Study to Investigate the Effects of CK-1827452 Injection on Ventricular Performance, Myocardial Oxygen Consumption, and Myocardial Efficiency in Patients With Heart Failure and Left Ventricular Systolic Dysfunction
Brief Title: Phase II Study of the Effect of CK-1827452 Injection on Myocardial Efficiency
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Decision to discontinue due to challenges of trial design and constraints on enrolling eligible and consenting patients.
Sponsor: Cytokinetics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CY 1124
Record Dates: First submitted 2008-04-21; First posted 2008-09-08 (Estimated); Results first posted 2010-08-23 (Estimated); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — omecamtiv mecarbil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort 1 (Experimental): 0.5 hour loading dose followed by 1.0 hour maintenance dose of CK-1827452
  Interventions: Drug: CK-1827452
- Cohort 2 (Experimental): ≤ 1.0 hour loading dose followed by 1.0 hour maintenance dose of CK-1827452
  Interventions: Drug: CK-1827452

INTERVENTIONS:
Drug: CK-1827452 — I.V. infusion for 0.5 hour at 54mg/hr followed by 1 hour at 21mg/hr
  Arms: Cohort 1
Drug: CK-1827452 — I.V. infusion for ≤ 1 hour at 72mg/hr followed by 1 hour at 36mg/hr
  Arms: Cohort 2

SUMMARY:
The purpose for this study (CY 1124) is to evaluate the effects of CK-1827452, a cardiac myosin activator, on myocardial systolic performance, myocardial oxygen consumption, and myocardial efficiency in patients with heart failure and to confirm that the unique preclinical pharmacological profile of CK- 1827452 is substantially the same in patients with heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Clinical indication for left and right heart catheterization
* Willing and able to provide informed consent
* Male or female 18 years of age or greater
* Symptomatic heart failure (≥ NYHA Class II)
* Ejection fraction ≤ 35%
* Patient is in sinus rhythm
* Patient is considered to be in suitable health in the opinion of the investigator, as determined by:

  o A pre-study physical examination with no clinical abnormalities which in the opinion of the investigator would preclude participation in the study other than physical symptoms or signs consistent with stable heart failure
* For female patients only: Post-menopausal or sterilized, or if she is of childbearing potential, she is not breastfeeding, her pregnancy test is negative, she has no intention to become pregnant for up to 90 days following the study, and she is using contraceptive drugs or devices

Exclusion Criteria:

* Acute myocarditis
* Hypertrophic, restrictive, or constrictive cardiomyopathy
* Congenital heart disease
* Known left ventricular thrombus
* Significant stenotic valvular disease (severe aortic stenosis, mitral stenosis)
* Poorly controlled hypertension (SBP > 180 mmHg)
* Pacemaker dependent ventricular rhythm
* Detectable troponin or CK-MB > ULN at any timepoint within 14 days of enrollment
* Acute coronary syndrome or revascularization procedure within 30 days of enrollment
* ≥ 50% stenosis of the left main coronary artery
* Plan for immediate revascularization procedure (PCI or CABG)
* GFR ≤ 35 ml/min/1.73 m2 by Modification of Diet in Renal Disease (MDRD) Equation or need for renal replacement therapy
* Known hepatic impairment (total bilirubin > 3 mg/dL, or ALT and AST > 2 times the upper limit of normal)
* Has received an investigational drug or device within 30 days before enrollment
* Has had any prior treatment with CK-1827452

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2008-09; Primary Completion 2008-11 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - Johns Hopkins Medical Institutions, Baltimore, Maryland
  - UUHSC / Division of Cardiology, Salt Lake City, Utah
- Mount Sinai Hospital, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period was from September 2008 to July 2009.
Groups:
- Mid Dose CK-1827452 (Cohort 1): 0.5 hour loading infusion followed by 1.0 hour maintenance infusion of CK-1827452
- High Dose CK-1827452 (Cohort 2): ≤ 1.0 hour loading infusion followed by 1.0 hour maintenance infusion of CK-1827452
Period: Overall Study
Arm/Group | Mid Dose CK-1827452 (Cohort 1) | High Dose CK-1827452 (Cohort 2)
Started | 2 | 0
Completed | 2 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Study was terminated due to challenges of trial design and constraints on enrolling eligible and consenting patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Mid Dose CK-1827452 (Cohort 1) | High Dose CK-1827452 (Cohort 2) | Total
Number analyzed (Participants) | 2 | 0 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 1 |  | 1
  >=65 years | 1 |  | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (13) |  | 69 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 |  | 2
  Male | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 |  | 2

OUTCOME MEASURES:

1. Primary Outcome: Effect of CK-1827452 on Myocardial Efficiency, Defined as the Ratio of Ventricular Performance to Myocardial Oxygen Consumption.
Description: Measure the effect CK-1827452 on hemodynamics and energetic measures of ventricular performance, myocardial oxygen consumption, and myocardial efficiency (the ratio of ventricular performance to myocardial oxygen consumption), in patients with clinical heart failure.
Time Frame: 1 day
Population: Study was terminated due to poor enrollment; 2 participants completed the study. Data quantity was insufficient to analyze or draw conclusions.
Arm/Group | Mid Dose CK-1827452 (Cohort 1) | High Dose CK-1827452 (Cohort 2)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Effects of CK-1827452 on Ventricular Performance
Description: Measure the effect of CK-1824752 on ventricular performance
Time Frame: 1 day
Population: No data displayed because Outcome Measure has zero total participants analyzed.
Arm/Group | Mid Dose CK-1827452 (Cohort 1) | High Dose CK-1827452 (Cohort 2)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Effects of CK-1827452 on Myocardial Oxygen Consumption
Description: Measure the effect of CK-1824752 on myocardial oxygen consumption
Time Frame: 1 day
Population: No data displayed because Outcome Measure has zero total participants analyzed.
Arm/Group | Mid Dose CK-1827452 (Cohort 1) | High Dose CK-1827452 (Cohort 2)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Effects of CK-1827452 on Pressure-volume Relationships
Description: Measure the effect of CK-1824752 on pressure-volume relationships
Time Frame: 1 day
Population: No data displayed because Outcome Measure has zero total participants analyzed.
Arm/Group | Mid Dose CK-1827452 (Cohort 1) | High Dose CK-1827452 (Cohort 2)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Effects of CK-1827452 on Systolic Ejection Time
Description: Measure the effect of CK-1824752 on systolic ejection time
Time Frame: 1 day
Population: No data displayed because Outcome Measure has zero total participants analyzed.
Arm/Group | Mid Dose CK-1827452 (Cohort 1) | High Dose CK-1827452 (Cohort 2)
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Effects of CK-1827452 on Invasively Measured Hemodynamics, Including Filling Pressure and Cardiac Output
Description: Measure the effect of CK-1824752 on invasively measured hemodynamics, including filling pressure and cardiac output
Time Frame: 1 day
Population: No data displayed because Outcome Measure has zero total participants analyzed.
Arm/Group | Mid Dose CK-1827452 (Cohort 1) | High Dose CK-1827452 (Cohort 2)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 30 days
Description: T
Arm/Group | Mid Dose CK-1827452 (Cohort 1) | High Dose CK-1827452 (Cohort 2)
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/0
Other Adverse Events (participants affected / at risk) | 2/2 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mid Dose CK-1827452 (Cohort 1) (N=2) | High Dose CK-1827452 (Cohort 2) (N=0)
Troponin Increased (Investigations) | 2 (2) | 0 (0) — The 2 troponin increases were mild in intensity and resolved.
Supraventricular Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) — The 1 supraventricular tachycardia was mild in intensity and resolved.

LIMITATIONS AND CAVEATS:
Inadequate enrollment led to early termination of study and insufficient number of patients for analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor's intention was to publish the results of the trial in collaboration with the Investigators.